CLINICAL TRIAL: NCT07404423
Title: Observational Prediction Model for Clinical Outcomes in Idiopathic Pulmonary Fibrosis: a Multicentre, ML-driven Study (OPEN-IPF)
Brief Title: OPEN-IPF: Observational Prediction modEl for cliNical Outcomes in Idiopathic Pulmonary Fibrosis
Acronym: OPEN-IPF
Status: Not yet recruiting | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Roberto Tonelli, MD, PhD, University of Modena and Reggio Emilia
Other Study IDs: UModenaReggio20262
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic pulmonary fibrosis; IPF; Disease progression; Acute exacerbation; Antifibrotic therapy; Nintedanib; Pirfenidone; Real-world data; Machine learning; Prognostic model; External validation; Multicentre cohort
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a progressive fibrotic lung disease with marked inter-individual heterogeneity in trajectories and outcomes. Despite antifibrotic therapies, reliable risk stratification in routine practice remains suboptimal. OPEN-IPF is a multicentre retrospective observational cohort study designed to build a harmonised real-world dataset across Italian IPF referral centres to enable the development and external validation of machine-learning (ML) models predicting clinically relevant outcomes.

DETAILED DESCRIPTION:
OPEN-IPF addresses the current limitation of AI/ML research in IPF-namely, the lack of large multicentre real-world datasets with harmonised variables and robust external validation. The study will retrospectively include adult patients with IPF followed in routine practice in participating Italian referral centres from 1 January 2015 to 31 December 2025 (data lock). No study-specific procedures will be performed. De-identified/pseudonymised data will be collected using a common data model, including demographics, smoking history, comorbidities, pulmonary function (FVC, DLCO), oxygen requirement, 6-minute walk test (where available), antifibrotic treatment exposure, HRCT features routinely reported, basic laboratory parameters, and clinical outcomes. The primary modelling targets are disease progression, acute exacerbations of IPF (AE-IPF), and real-world response to antifibrotic treatment. Model development will be performed using multicentre data with explicit external validation across centres

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of idiopathic pulmonary fibrosis established according to international guidelines and local multidisciplinary team (MDT) assessment
* Availability of baseline clinical and functional data
* Availability of follow-up data for at least 12 months, or until a clinically relevant event (e.g., death, lung transplantation)

Exclusion Criteria:

* Interstitial lung disease other than IPF
* Lung transplantation performed before the baseline (index) date
* Absence of any follow-up information after baseline

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with idiopathic pulmonary fibrosis diagnosed according to international guidelines and local multidisciplinary team assessment, followed in routine care at participating Italian referral centres.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Disease progression (guideline-based functional/composite criteria) | From baseline (index date) up to 12 months and up to end of available follow-up (maximum: 31 December 2025)
  Disease progression defined using guideline-based criteria derived from routinely collected clinical data (e.g., decline in lung function and/or composite progression definitions as per the shared operational document).

SECONDARY OUTCOMES:
Acute exacerbation of IPF (AE-IPF) | From baseline to end of follow-up (maximum: 31 December 2025)
  Occurrence of AE-IPF during follow-up, adjudicated from routine clinical documentation using standardised operational definitions shared across centres.
Real-world response to antifibrotic therapy | From treatment initiation (or baseline if already treated) up to 12 months and end of follow-up (maximum: 31 December 2025)
  Treatment response assessed in routine clinical practice using longitudinal clinical/functional data and treatment exposure information (type, start, discontinuation)
Overall survival | From baseline to end of follow-up (maximum: 31 December 2025)
  Time from baseline to death from any cause.
Transplant-free survival | From baseline to end of follow-up (maximum: 31 December 2025)
  Time from baseline to lung transplantation or death.
Time to first progression or AE-IPF event | From baseline to end of follow-up (maximum: 31 December 2025)
  Time from baseline to first occurrence of disease progression or AE-IPF.

IPD SHARING:
Plan to Share IPD: Undecided